CLINICAL TRIAL: NCT01160354
Title: Phase I/II Study of Plerixafor and Clofarabine in Previously Untreated Older (>/=60 Years) Adult Patients With Acute Myelogenous Leukemia (AML) With Two or More Unfavorable Prognostic Factors for Whom Standard Induction Chemotherapy is Unlikely to be of Benefit
Brief Title: Plerixafor and Clofarabine in Frontline Treatment of Elderly Patients With Acute Myelogenous Leukemia (AML)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0536; NCI-2012-01786 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Leukemia; AML; Clofarabine; Plerixafor; elderly patients; previously untreated; unfavorable prognostic factors
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — plerixafor; Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plerixafor 240 mcg/kg + Clofarabine (Experimental): Plerixafor 240 mcg/kg daily subcutaneous (SQ) injection on Days 1-5, 4-6 hours before hour IV administration of Clofarabine fixed dose of 30 mg/m2/day during Induction cycle (20 mg/m2/day in consolidation cycles).
  Phase II: Plerixafor at the highest dose tolerated in Phase I.
  Plerixafor was dose-escalated in a 3+3 design, starting at 240 mcg/kg, and proceeding to dose levels of 320 mcg/kg, and 400 mcg/kg.
  Interventions: Drug: Plerixafor; Drug: Clofarabine

INTERVENTIONS:
Drug: Plerixafor — Starting at 240 mcg/kg daily subcutaneous (SQ) injection on Days 1-5, 4-6 hours before a 1 hour (+/- 30 minutes) IV administration of Clofarabine
  Other Names: Mobozil
Drug: Clofarabine — Fixed dose of 30 mg/m2/day during Induction cycle (20 mg/m2/day in consolidation cycles).
  Other Names: Clofarex; Clolar

SUMMARY:
The goal of Part 1 of this clinical research study is to learn about the safety of the combination of plerixafor and clofarabine when given to patients with previously untreated AML who are at least 60 years old.

The goal of Part 2 of this study is to learn if the combination of plerixafor and clofarabine can help to control previously untreated AML in patients who are at least 60 years old. Study was closed early and did not progress to Part 2.

DETAILED DESCRIPTION:
The Study Drugs:

Plerixafor is designed to block a protein on cancer cells from attaching to cells in the bone marrow. This may allow cells in the bone marrow to be more effectively treated by chemotherapy.

Clofarabine is designed to interfere with the growth and development of cancer cells.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. Up to 3 groups of up to 6 participants will be enrolled in the Part 1 portion of the study, and up to 48 participants will be enrolled in Part 2.

If you are enrolled in Part 1, the dose of plerixafor you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of plerixafor. Each new group will receive a higher dose of plerixafor than the group before it, if no intolerable side effects were seen.

If you are enrolled in Part 2, you will receive plerixafor at the highest dose that was tolerated in Part 1.

All participants will receive the same doses of clofarabine.

Study Drug Administration:

Cycles in this study are 28 days long, or possibly longer depending on your blood counts, any side effects, and the status of the disease.

On Days 1-5 of each cycle, you will receive plerixafor through a needle under the skin of your abdomen.

On Days 1-5 of each cycle, you will receive clofarabine by vein over about 1 hour. The dose will begin about 4 to 6 hours after the plerixafor injection. You will be watched for side effects while you receive clofarabine.

If the doctor thinks it is in your best interest, the dose level of plerixafor may be lowered.

Cycle 1 is called Induction. If the disease goes into remission (responds well) after the Induction cycle, you will start the Consolidation part of the study. In the Consolidation cycles, the schedule of administration of the drugs will be the same as in the Induction cycle, but the doses of clofarabine will be lower. If the disease does not go into remission after the Induction cycle, you will have a Reinduction cycle before you can begin the Consolidation part of the study. The goal of the Induction cycle and possible Reinduction cycle is to affect the bone marrow a certain way that may help control the disease. The goal of Consolidation is also to help control the disease.

Study Visits:

Induction (Cycle 1):

On Day 1 of Induction, blood (about ½ tablespoon each time) will be drawn for routine tests before the plerixafor injection and 3 times during the 8 hours after the injection.

On Days 2-5 of Induction, blood (about ½ tablespoon each time) will be drawn for routine tests before the plerixafor injection and again at 8 hours after the injection.

Starting in Week 2 of Induction, blood (about 2 tablespoons) will be drawn at least 2 times a week for routine tests.

You will have a bone marrow aspiration and/or biopsy to check the status of the disease on Day 21 of Induction and every 2 weeks after that, until the Induction cycle is over.

Reinduction:

If you have a Reinduction cycle, blood (about 2 tablespoons) will be drawn at least 2 times a week during Reinduction for routine tests. You will have a bone marrow aspiration and/or biopsy to check the status of the disease on Day 21 of Reinduction and every 2 weeks after that, until the Reinduction cycle is over.

Consolidation:

Blood (about 2 tablespoons) will be drawn 1 time a day for routine tests on Days 1-5 of Consolidation.

Starting in Week 2 of each Consolidation cycle, blood (about 2 tablespoons) will be drawn for routine tests every week for the rest of each Consolidation cycle.

You will have a bone marrow aspiration and/or biopsy to check the status of the disease anytime during Consolidation that the doctor decides it is needed.

Induction, Reinduction, and Consolidation:

The blood tests and/or bone marrow aspirations/biopsies may be performed more often than listed if the doctor thinks it is needed. Also, you will have an ECG anytime during the study if the doctor thinks it is needed.

Length of Study:

You may continue taking the study drugs for up to 5 Consolidation cycles, if the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse or intolerable side effects occur.

Your participation on the study will be over once you have completed the follow-up visits.

Follow-Up Visits:

At 1 and 3 months after you stop taking the study drugs:

* Blood (about 2 tablespoon) will be drawn for routine tests.
* If the doctor decides it is needed, you will have a bone marrow aspiration to check the status of the disease.

If the disease responds (if it goes into complete or partial remission), you will have follow-up visits every 3 months for up to 2 years after you stop taking the study drugs. The follow-up visits will stop if the disease gets worse, or if you start a new cancer therapy and the disease has not gotten worse. The following tests and procedures will be performed at the follow-up visits:

* Blood (about 2 tablespoon) will be drawn for routine tests.
* If the doctor decides it is needed, you will have a bone marrow aspiration to check the status of the disease.

This is an investigational study. Clofarabine is FDA approved and commercially available to treat acute lymphoblastic leukemia (ALL) in children after the disease has gotten worse a second time. Plerixafor is FDA approved to be given with G-CSF and is commercially available for use in moving stem cells into the bloodstream before a stem cell transplant to treat non-Hodgkin's lymphoma or multiple myeloma. The combination of clofarabine and plerixafor is investigational.

Up to 66 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 60 years
2. Diagnosis of untreated AML (de novo, secondary, or with an antecedent hematologic disorder [AHD]) according to the World Health Organization (WHO) criteria
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
4. At least 2 of the following adverse prognostic factors: Age >/= 70 years; or AHD; or ECOG performance status of = 2; or intermediate or unfavorable (ie, adverse) karyotype defined as any cytogenetic profile except the presence of any of the following: t(8;21)(q22;q22), inv(16)(p13q22) or t(16;16)(p13;q22), t(15;17)(q22;q12) and variants.
5. Provide signed, written informed consent.
6. Be able to comply with study procedures and follow-up examinations.
7. Adequate renal and hepatic function as indicated by all of the following: Total bilirubin </=1.5 x institutional Upper Limit of Normal (ULN); an Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) </=2.5 x Upper limits of normal (ULN); and an estimated creatinine clearance (CrCl) of > 50 mL/min, as calculated by the Cockcroft -Gault equation.
8. Adequate cardiac function as measured by at least 1 of the following: Left ventricular ejection fraction (LVEF) >/=40% on multigated acquisition (MUGA) scan or similar radionuclide angiographic scan; or Left ventricular fractional fractional shortening >/=22% on echocardiography exam; or LVEF >/=40% on echocardiography exam.
9. Women of child-bearing potential (WOCBP) must agree to use adequate birth control through the end of the last treatment visit. WOCBP is a women who has not been naturally postmenopausal for at least 12 consecutive months or who had not undergone previous surgical sterilization.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL), (French-American-British classification M3 or WHO classification of APL with t(15;17)(q22;q12), (PML/RAR alpha fusion gene and variants).
2. Prior treatment with clofarabine.
3. Prior treatment for AML or an AHD (excluding supportive care, hydroxyurea, hematopoietic cytokines, or lenalidomide [the latter specifically for an AHD only]). Hematopoietic cytokines and lenalidomide must not have been received within 14 days prior to first dose of study drug; hydroxyurea is allowed on study to control white blood cell count (WBC) counts. If any of the above treatments have been received for AML or an AHD within the permissible time periods, drug-related toxicities must have recovered to Grade 1 or less prior to first dose of study drug.
4. Prior hematopoietic stem cell transplant (HSCT).
5. Prior external beam radiation therapy to the pelvis.
6. Investigational agent received within 30 days prior to the first dose of study drug. If received any investigational agent prior to this time point, drug-related toxicities must have recovered to Grade 1 or less prior to first dose of study drug.
7. Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
8. Any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo therapy with clofarabine.
9. Clinical evidence suggestive of central nervous system (CNS) involvement with leukemia unless a lumbar puncture confirms the absence of leukemic blasts in the cerebrospinal fluid (CSF)
10. Prior positive test for the human immunodeficiency virus (HIV).
11. WBC >50 × 10^9/L; the first 3 patients enrolled on the study will be required to have a WBC of <20 × 10^9/L.
12. Have psychiatric disorders that would interfere with consent, study participation, or follow-up.
13. Have been diagnosed with another malignancy, unless the patient has been disease free for at least 5 years following curative intent therapy, following exceptions: Patients with treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of disease-free duration, if definitive treatment for the condition has been completed or patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values if hormonal therapy has been initiated or radical prostatectomy has been performed.
14. Are pregnant or lactating.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan A. Burger, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 05, 2010 to May 13, 2014. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Study was closed early due to slow accrual and did not continue to complete second part (Phase 2). Last cohort of Maximum Tolerated Dose (MTD) level 400 mgc/kg included two participant registrations for study continuation that did not occur.
Groups:
- Plerixafor 240 mcg/kg + Clofarabine: Plerixafor 240 mcg/kg daily subcutaneous (SQ) injection on Days 1-5, 4-6 hours before hour intravenous (IV) administration of Clofarabine fixed dose of 30 mg/m2/day during Induction cycle (20 mg/m2/day in consolidation cycles).
- Plerixafor 320 mcg/kg + Clofarabine: Plerixafor 320 mcg/kg daily SQ injection on Days 1-5, 4-6 hours before hour IV administration of Clofarabine fixed dose of 30 mg/m2/day during Induction cycle (20 mg/m2/day in consolidation cycles).
- Plerixafor 400 mcg/kg + Clofarabine: Plerixafor 400 mcg/kg daily SQ injection on Days 1-5, 4-6 hours before hour IV administration of Clofarabine fixed dose of 30 mg/m2/day during Induction cycle (20 mg/m2/day in consolidation cycles).
Period: Overall Study
Arm/Group | Plerixafor 240 mcg/kg + Clofarabine | Plerixafor 320 mcg/kg + Clofarabine | Plerixafor 400 mcg/kg + Clofarabine
Started | 3 | 4 | 15
Completed | 3 | 3 | 14
Not Completed | 0 | 1 | 1
Not completed — Death | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Plerixafor 240 mcg/kg + Clofarabine: Plerixafor 240 mcg/kg daily subcutaneous (SQ) injection on Days 1-5, 4-6 hours before hour IV administration of Clofarabine fixed dose of 30 mg/m2/day during Induction cycle (20 mg/m2/day in consolidation cycles).
- Total: Total of all reporting groups
Arm/Group | Plerixafor 240 mcg/kg + Clofarabine | Plerixafor 320 mcg/kg + Clofarabine | Plerixafor 400 mcg/kg + Clofarabine | Total
Number analyzed (Participants) | 3 | 4 | 15 | 22
Age, Continuous [Median (Full Range); unit: years] | 69 [67 to 76] | 69 [66 to 72] | 72 [61 to 81] | 71 [61 to 81]
Age, Customized [Count of Participants; unit: Participants]
  Range of Years: 60-69 | 2 | 2 | 4 | 8
  Range of Years: 70-79 | 1 | 2 | 10 | 13
  Range of Years: 80+ | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 5 | 9
  Male | 2 | 1 | 10 | 13
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 15 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Phase I With First Cycle Dose Limiting Toxicities (DLT) Observed
Description: Dose limiting toxicity (DLT) consists of participants who developed DLT during maximum tolerated dose (MTD) estimation period where DLTs observed during dose escalation were used to develop MTD. The MTD is the highest dose level in which <2 participants of 6 develop first cycle. DLT. Toxicity graded according to the NCI Common Toxicity Criteria Version 3.0. The timeframe to assess dose-limiting toxicities (DLT's) will be the first cycle of treatment, i.e. the first 4 weeks on study. The Plerixafor dose to be used in Phase II of the protocol is the highest dose at which no more than 1 of 6 patients experience a DLT in the Phase I part of the protocol or a lower dose selected at the end of dose escalation.
Time Frame: First cycle of treatment, i.e. first 4 weeks on study
Population: Intent to treat population included all registered participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Plerixafor 240 mcg/kg + Clofarabine | Plerixafor 320 mcg/kg + Clofarabine | Plerixafor 400 mcg/kg + Clofarabine
Number analyzed (Participants) | 3 | 4 | 15
Participants | 0 | 0 | 0

2. Secondary Outcome: Participants' Response During First Part of Study
Description: Response defined as Complete remission (CR): Disappearance all clinical +/or radiologic evidence disease. Neutrophil count >/=1.0x10^9/L & platelet count >/=100x10^9/L, & normal bone marrow differential (</= 5% blasts). Complete Remission without Platelet Recovery (CRp): Peripheral blood & bone marrow results as for CR, but with platelet counts of <100x10^9/L. Partial Remission (PR): Blood count recovery as for CR, but both decrease in marrow blasts >50% & not more than 6 to 25% abnormal cells in the marrow.
Time Frame: Assessments following 3 cycles (at 12 weeks) up to 5 cycles (20 weeks)
Population: Two participants were not evaluable due to unrelated early death.
Measure: Count of Participants; unit: Participants
Arm/Group | Plerixafor 240 mcg/kg + Clofarabine | Plerixafor 320 mcg/kg + Clofarabine | Plerixafor 400 mcg/kg + Clofarabine
Number analyzed (Participants) | 3 | 3 | 14
Participants
  CR | 2 | 1 | 5
  CRp | 0 | 0 | 3
  PR | 0 | 0 | 1
  Marrow CR | 0 | 0 | 2
  No Response, Resistant | 1 | 2 | 3

3. Secondary Outcome: Number of Participants With Overall Response During Second Part of Study
Description: Overall response (OR) = Complete Remission (CR) + Partial Remission (PR) where response defined: Complete remission (CR): Disappearance all clinical +/or radiologic evidence disease. Neutrophil count >/=1.0x109/L & platelet count >/=100x10^9/L, & normal bone marrow differential (</= 5% blasts). Complete Remission without Platelet Recovery (CRp): Peripheral blood & bone marrow results as for CR, but with platelet counts of <100x10^9/L. Partial Remission (PR): Blood count recovery as for CR, but both decrease in marrow blasts >50% & not more than 6 to 25% abnormal cells in the marrow. Treatment Failure: For purposes of efficacy analysis of remission, less than a CR, CRi, or PR categorized as Treatment Failure.
Time Frame: Continuously monitored, assessments at 12 weeks
Population: Study halted early without continuing to second part (Phase II). This outcome measure is to analyze the overall response during the Phase II portion of this study. The study was halted early and did not enroll any patients in the phase II portion. Therefore, there are Zero patients to analyze and no data to report.
Arm/Group | Plerixafor 240 mcg/kg + Clofarabine | Plerixafor 320 mcg/kg + Clofarabine | Plerixafor 400 mcg/kg + Clofarabine
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collected during 28-day cycle, up to 6 cycles (24 weeks).
Arm/Group | Plerixafor 240 mcg/kg + Clofarabine | Plerixafor 320 mcg/kg + Clofarabine | Plerixafor 400 mcg/kg + Clofarabine
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/4 | 1/15
Serious Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 15/15
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plerixafor 240 mcg/kg + Clofarabine (N=3) | Plerixafor 320 mcg/kg + Clofarabine (N=4) | Plerixafor 400 mcg/kg + Clofarabine (N=15)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Angina (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrilation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Elevated alanine aminotransferase (ALT (Investigations) | 0 (0) | 0 (0) | 1 (1)
Elevated Renal Function (creatinine) (Investigations) | 0 (0) | 0 (0) | 1 (1)
Elevated renal function (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fungal Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection Blood (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenic fever (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 6 (11)
Oral Herpes Simplex Virus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Prolonged Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plerixafor 240 mcg/kg + Clofarabine (N=3) | Plerixafor 320 mcg/kg + Clofarabine (N=4) | Plerixafor 400 mcg/kg + Clofarabine (N=15)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5) | 5 (6)
Increased Alanine aminotransferase (ALT) (Investigations) | 3 (4) | 2 (3) | 4 (9)
Increased Aspartate aminotransferase (AST) (Investigations) | 0 (0) | 0 (0) | 1 (1)
Increased bilirubin (Investigations) | 1 (2) | 0 (0) | 5 (5)
Constiptation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Increased creatinine (Investigations) | 1 (1) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Increased Lipase (Investigations) | 0 (0) | 0 (0) | 1 (2)
Nausea (General disorders) | 2 (3) | 2 (2) | 10 (21)
Neuropathy - Sensory (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Other than general (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 6 (11)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination led to no subjects analyzed for later period outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes